CLINICAL TRIAL: NCT02676791
Title: Influence of Esophageal Washout on Local Carcinoma Recurrence After Curative Resection - a Randomized Controlled Trial
Brief Title: Influence of Esophageal Washout on Local Carcinoma Recurrence After Curative Resection
Acronym: LOCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VTG-07
Record Dates: First submitted 2016-02-04; First posted 2016-02-08 (Estimated); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Povidone-Iodine) (Experimental): Esophageal washout will be performed via a nasogastric tube with approx. 50ml of a 11% povidone-iodine solution (Betaisodona®, Mundipharma) during esophageal resection.
  Interventions: Drug: Povidone-Iodine
- B (Control) (No Intervention): Esophageal resection will be performed without esophageal washout.

INTERVENTIONS:
Drug: Povidone-Iodine — A standard nasogastric tube will be inserted into all patients after induction of general anesthesia. After surgical dissection, the esophagus / stomach will be cut at the desired level leaving the tip of the nasogastric tube proximal to the esophageal carcinoma. Then, 50ml of a 11% povidone-iodine solution (Betaisodona®, Mundipharma) will be introduced into the esophagus via the nasogastric tube and evacuated with a suction device (washout). The nasogastric tube will then be removed for completion of esophageal resection and beginning of reconstruction.
  Other Names: Betaisodona
  Arms: A (Povidone-Iodine)

SUMMARY:
The LOCARE-Trial is an investigator initiated, randomized-controlled trial with two parallel arms (n=60 each) and investigates the influence of esophageal washout on long-term outcomes in patients undergoing elective esophageal resection for carcinoma. The primary endpoint is defined as local carcinoma recurrence. Secondary endpoints will be locoregional and distant recurrence, disease-specific survival and esophageal cancer specific survival.

DETAILED DESCRIPTION:
Treatment of squamous cell carcinoma and adenocarcinoma of the esophagus has changed rapidly over the last decades due to implementation of multimodal cancer therapies such as radiotherapy or combined radiochemotherapy. Surgery, however, still is the mainstay of curative treatment options for this cancer entity. Due to the significant improvement in surgical technique and perioperative management, the postoperative mortality rate has fallen to about 5% with an estimated 5-year survival of 35%. Nevertheless, patients after esophagectomy are at high risk for local recurrence especially within the first 2 years after treatment. Independent risk factors for the development of carcinoma recurrence are incomplete resection (R1), extracapsular lymph node involvement and postoperative complications. Exfoliated, malignant cells remaining in luminal organs like the esophagus or colorectum could present another important risk factor for local recurrence especially at the site of anastomosis. In the treatment of rectal cancer, data have shown, that intraoperative rectal washout significantly reduces the risk of local recurrence from about 10% to 5%. For this reason, rectal washout during anterior resection has become a standard in many surgical institutions. Besides agents like cetrimide, sodium hypochlorite, formalin or saline, povidone-iodine has also been used for rectal mucosal application in prospective studies. Questions arise, weather similar positive outcomes could be achieved in esophageal surgery. The investigators hypothesize that esophageal washout with a povidone-iodine solution (Betaisodona®, Mundipharma) reduces the risk of local carcinoma recurrence after radical resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective esophageal resection or esophagectomy
* Age equal or greater than 18 years
* Written informed consent
* Squamous cell carcinoma of the esophagus (SCC)
* Adenocarcinoma of the gastroesophageal junction (AEG) Type I

Exclusion Criteria:

* Local irresectability or metastatic disease
* Adenocarcinoma of the gastroesophageal junction Type II and III
* Histopathological R1-resection
* Surgery for recurrence
* Iodine allergy
* Hyperthyreosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Local carcinoma recurrence | 36 months
  Defined as development of a local recurrence after surgical treatment for esophageal cancer. The tumor is of identical histopathological type and occurs either on remained parts of the esophagus, at the site of anastomosis, on parts of an interposed organ (i.e. jejunum or colon) or in the original esophageal bed.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Reißfelder, MD, Principal Investigator — Department of GI, Thoracic and Vascular Surgery, University Hospital Carl Gustav Carus, TU Dresden
Locations (1):
- Department of GI, Thoracic and Vascular Surgery, University Hospital Carl Gustav Carus, TU Dresden, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No